CLINICAL TRIAL: NCT06093334
Title: iMagINg of Chemotherapy-Induced Morphological and Functional Lung Changes in Childhood Acute Lymphoblastic Leukemia and Hodgkin's Disease
Brief Title: Imaging of Chemotherapy-induced Morphological and Functional Lung Changes in Childhood ALL and HD
Acronym: MinimALL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-47-B
Record Dates: First submitted 2023-10-04; First posted 2023-10-23 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Acute Lymphoblastic Leukemia; Hodgkin Disease; Allogeneic Stem Cell Transplantation
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease | interventions — Exercise Test; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early therapeutic effects (Experimental): Diagnosed acute lymphatic leukemia or Hodgkin's disease (HD) and completed induction therapy or radiotherapy, from 5 years to <18 years
  Interventions: Diagnostic Test: Low-field magnetic resonance imaging; Diagnostic Test: Cardiopulmonary testing; Diagnostic Test: Pulmonary testing; Diagnostic Test: Blood sample
- Late therapeutic effects (Experimental): Diagnosed acute lymphatic leukemia or Hodgkin's disease (HD) and completed intensive therapy or radiotherapy, Patient in follow-up care, from 5 years to <18 years
  Interventions: Diagnostic Test: Low-field magnetic resonance imaging; Diagnostic Test: Cardiopulmonary testing; Diagnostic Test: Pulmonary testing; Diagnostic Test: Blood sample
- Effects of hematopoietic stem cell transplantation (Experimental): Diagnosed acute lymphatic leukemia, completed hematopoietic stem cell transplantation, from 5 years to <18 years
  Interventions: Diagnostic Test: Low-field magnetic resonance imaging; Diagnostic Test: Cardiopulmonary testing; Diagnostic Test: Pulmonary testing; Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Low-field magnetic resonance imaging — Imaging of lung parenchyma and function by LF-MRI
Diagnostic Test: Cardiopulmonary testing — Myocardial function (Strain-Analysis by echocardiography) and spiroergometry, capillary blood gases and lactate
Diagnostic Test: Pulmonary testing — Lung function (VC%, FEV1%)
Diagnostic Test: Blood sample — Standard procedures/parameters routinely available in follow-up care after oncological treatment

SUMMARY:
With increasing cure rates of childhood cancer there is growing recognition of late effects of treatments. However, there is a lack of non-invasive and child-friendly procedures that can indicate possible late damage. This study uses morphologic and free-breathing phase-resolved functional low-field (PREFUL) magnetic resonance imaging (MRI) to identify persistent pulmonary toxicity after treatment for childhood acute lymphoblastic leukemia (ALL), Hodgkin's disease (HD) and allogeneic stem cell transplantation. Furthermore, cardiopulmonary testing is performed by means of a pulmonary function test, echocardiography with strain analysis and spiroergometry.

DETAILED DESCRIPTION:
With increasing cure rates of childhood cancer there is growing recognition of late effects of treatments. However, there is a lack of non-invasive and child-friendly procedures that can indicate possible late damage.

This study uses morphologic and free-breathing phase-resolved functional low-field (PREFUL) magnetic resonance imaging (MRI) to identify persistent pulmonary toxicity after treatment for childhood acute lymphoblastic leukemia (ALL), Hodgkin's disease (HD) and allogeneic stem cell transplantation. The examination in the new 0.55 T MRI system does not differ in procedure and especially with regard to contraindications for an MRI examination from an examination in routinely used 1.5 or 3T devices. There is no intravenous administration of contrast medium. This method has already yielded relevant results in a previous study on the frequency of lung parenchymal changes in pediatric and adolescent patients with past SARS-CoV-2 infection detected by PCR. In addition, study participants will undergo cardiopilmonary testing by spirometry, spiroergometry and echocardiography with strain analysis to assess cardiac and pulmonary performance. For the individual patient, the duration of study participation is 120 minutes. This includes approximately 30 minutes for education and consent of study participants/parents/guardians, 30 minutes for lung function test and MRI, and 30 minutes for cardiopulmonary testing.

The purpose of this study is to assess early posttherapeutic changes as well as possible persistent pulmonary toxicity and change in cardiopulmonary performance.

ELIGIBILITY:
Study arm: "Early therapeutic effects"

Inclusion Criteria:

* Diagnosed acute lymphatic leukemia or Hodgkin's disease (HD)
* Completed induction therapy or radiotherapy

Exclusion Criteria:

* Pregnancy, Lactation
* Known pleural or pericardial effusion
* Critical condition (requiring respiratory support, ventilation, oxygen, shock, symptomatic heart failure)
* Marked thoracic deformities/malformations
* Previous lung surgery
* Injuries that do not allow physical stress diagnostics
* Rejection of MRI imaging
* General contraindications for MRI examinations (e.g. electrical implants such as cardiac pacemakers or perfusion pumps, etc.)

Study arm: "Late therapeutic effects"

Inclusion Criteria:

* Diagnosed acute lymphatic leukemia or Hodgkin's disease (HD)
* Completed intensive therapy or radiotherapy

Exclusion Criteria:

* Pregnancy, Lactation
* Known pleural or pericardial effusion
* Critical condition (requiring respiratory support, ventilation, oxygen, shock, symptomatic heart failure)
* Marked thoracic deformities/malformations
* Previous lung surgery
* Injuries that do not allow physical stress diagnostics
* Rejection of MRI imaging
* General contraindications for MRI examinations (e.g. electrical implants such as cardiac pacemakers or perfusion pumps, etc.)

Study arm: "Effects of hematopoietic stem cell transplantation"

Inclusion Criteria:

* Diagnosed acute lymphatic leukemia
* Completed hematopoietic stem cell transplantation

Exclusion Criteria:

* Pregnancy, Lactation
* Known pleural or pericardial effusion
* Critical condition (requiring respiratory support, ventilation, oxygen, shock, symptomatic heart failure)
* Marked thoracic deformities/malformations
* Previous lung surgery
* Injuries that do not allow physical stress diagnostics
* Rejection of MRI imaging
* General contraindications for MRI examinations (e.g. electrical implants such as cardiac pacemakers or perfusion pumps, etc.)

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Morphologic lung assessment (LF-MRI) | Single time point (1 day)
  Morphologic changes in lung parenchyma

SECONDARY OUTCOMES:
Functional lung assessment (LF-MRI) | Single time point (1 day)
  Change in functional lung parameters
Cardiopulmonary testing (VO2) | Single time point (1 day)
  Oxygen uptake
Cardiopulmonary testing (VO2max) | Single time point (1 day)
  Peak oxygen uptake
Cardiopulmonary testing (RER) | Single time point (1 day)
  Respiratory exchange ratio
Cardiopulmonary testing (VT2) | Single time point (1 day)
  Ventilatory anaerobic threshold
Cardiopulmonary testing (VCO2) | Single time point (1 day)
  Carbon dioxide output
Cardiopulmonary testing (HR) | Single time point (1 day)
  Heart rate
Cardiopulmonary testing (HRR) | Single time point (1 day)
  Heart Rate Reserve
Cardiopulmonary testing (Breath rate at VAT) | Single time point (1 day)
  Breath rate at VAT
Cardiopulmonary testing (BRR) | Single time point (1 day)
  Breath rate reserve
Cardiopulmonary testing (VE) | Single time point (1 day)
  Minute Ventilation
Cardiopulmonary testing (O2-Pulse) | Single time point (1 day)
  O2-Pulse
Cardiopulmonary testing (HRV) | Single time point (1 day)
  Heart rate variability
Cardiopulmonary testing (Borg-Scale) | Single time point (1 day)
  Exercise capacity (Borg-Scale)
Cardiopulmonary testing (VO2) | Single time point (1 day)
  Capillary blood gases and lactate
Cardiopulmonary testing (Strain-Analysis) | Single time point (1 day)
  Strain-Analysis by echocardiography
Pulmonary test (Lung function) | Single time point (1 day)
  Lung function (VC%, FEV1%)
Blood sample (Blood count) | Single time point (1 day)
  Blood Count
Blood sample (Enterocytes) | Single time point (1 day)
  Concentration of Enterocytes
Blood sample (Liver enzymes) | Single time point (1 day)
  Liver enzymes
Blood sample (Retention parameters) | Single time point (1 day)
  Concentration of kreatinin and urea
Weight | Single time point (1 day)
  Weight of the participant in kilograms
Height | Single time point (1 day)
  Height of the participant in meters

CONTACTS AND LOCATIONS:
Overall Officials: Axel Karow, MD, Principal Investigator — Department of Pediatrics and Adolescent Medicine, University Hospital Erlangen; Ferdinand Knieling, MD, Principal Investigator — Department of Pediatrics and Adolescent Medicine, University Hospital Erlangen; Rafael Heiß, MD, Principal Investigator — Institute of Radiology, University Hospital Erlangen
Locations (1):
- Department of Pediatrics and Adolescent Medicine, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request as follows:
  Individual participant data will not be available Study Protocol and Statistical Analysis Plan will be available The data will be available beginning 9 months and ending 36 months following article publication.
  The data will be available to researchers who provide a methodologically sound proposal.
  The data will be available for individual participant data meta-analysis, only. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at https://www.uk-erlangen.de.
  Restrictions may apply due to patient privacy and the General Data Protection Regulation.

REFERENCES:
- [Background] Erdmann F, Frederiksen LE, Bonaventure A, Mader L, Hasle H, Robison LL, Winther JF. Childhood cancer: Survival, treatment modalities, late effects and improvements over time. Cancer Epidemiol. 2021 Apr;71(Pt B):101733. doi: 10.1016/j.canep.2020.101733. Epub 2020 May 24. PMID 32461035
- [Background] Silverman LB. Balancing cure and long-term risks in acute lymphoblastic leukemia. Hematology Am Soc Hematol Educ Program. 2014 Dec 5;2014(1):190-7. doi: 10.1182/asheducation-2014.1.190. Epub 2014 Nov 18. PMID 25696854
- [Background] Gebauer J, Baust K, Bardi E, Grabow D, Stein A, van der Pal HJ, Calaminus G, Langer T. Guidelines for Long-Term Follow-Up after Childhood Cancer: Practical Implications for the Daily Work. Oncol Res Treat. 2020;43(3):61-69. doi: 10.1159/000504200. Epub 2020 Jan 13. PMID 31931503
- [Derived] Huber F, Schoeffl I, Mueller N, Dierl A, Wild EM, Naumann-Bartsch N, Karow A, Knieling F, Woelfle J, Dittrich S, Anderheiden F. What about the heart - pediatric ALL survivors show cardiopulmonary limitations in the MinimALL Study. Eur J Pediatr. 2025 Jun 9;184(7):406. doi: 10.1007/s00431-025-06243-0. PMID 40488780

DOCUMENTS (2):
  • Study Protocol (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT06093334/Prot_002.pdf
  • Statistical Analysis Plan (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT06093334/SAP_003.pdf